CLINICAL TRIAL: NCT03187106
Title: Prophylactic Antibiotics After Cesarean
Acronym: PACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 17-0035
Record Dates: First submitted 2017-06-12; First posted 2017-06-14 (Actual); Last update posted 2023-08-16 (Actual); Status verified 2023-08

CONDITIONS: Surgical Site Infection
MeSH Terms: conditions — Surgical Wound Infection | interventions — Cephalexin; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Cephalexin and metronidazole (Experimental): 500 mg cephalexin per oral every 8 hours for a total of 6 doses; 500 mg metronidazole per oral every 8 hours for a total of 6 doses
  Interventions: Drug: Cephalexin; Drug: Metronidazole
- Placebo / standard of care (Placebo Comparator): Placebo pills per oral every 8 hours for a total of 6 doses
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Cephalexin — Other name(s): Keflex (cephalexin) Cephalexin at 500 mg per oral every 8 hours for a total of 6 doses
  Arms: Cephalexin and metronidazole
Drug: Placebo — Placebo representing standard of care
  Arms: Placebo / standard of care
Drug: Metronidazole — Other name(s): Flagyl (metronidazole) Metronidazole at 500 mg per oral every 8 hours for a total of 6 doses
  Arms: Cephalexin and metronidazole

SUMMARY:
The purpose of this study is to determine if the addition of a 48-hour course of post-operative antibiotics to the recommended course of pre-operative antibiotics improves surgical site infection rate in patients who are obese and undergo Cesarean section after laboring.

DETAILED DESCRIPTION:
The investigators propose the conduction of a prospective, randomized, double-blinded clinical trial to evaluate an alternative prophylactic regimen for the prevention of surgical site infection in women who are obese and have been laboring prior to their Cesarean section. This study is to be conducted by the Department of Obstetrics & Gynecology at John Sealy Hospital at the University of Texas Medical Branch in Galveston, Texas. The intervention being studied will be the administration of cephalexin and metronidazole post-operatively for 48 hours. The primary outcome measure will be surgical site infection (including superficial or deep incisional surgical site infection, endometritis, and other related infections, such as septic pelvic thrombophlebitis and abdominal or pelvic abscess) in the post-operative period.

In order to most effectively and accurately analyze our primary and secondary research outcomes, the investigators will standardize our surgical operation techniques in all ways feasible. These recommendations will be in concordance with American College of Obstetrics and Gynecology recommendations, as those generally accepted in the medical literature. All patients will undergo surgery in the same small group of HEPA-filtered and positive air-pressure operating rooms. Appropriate limitations on number of surgeons and assistants scrubbed for surgery, as well as general OR traffic, will be enforced. Patients will undergo hair clipping of the incision site when appropriate. Chlorhexidine skin decontamination will be the standard surgical site preparation. An adhesive drape will be used. Prior to skin incision, cefazolin and azithromycin will be administered.

All patients to be considered for recruitment to this study will be undergoing delivery at John Sealy Hospital at the University of Texas Medical Branch in Galveston, Texas. Patients with an elevated BMI >or =30 kg/m2 who undergo cesarean section after laboring will be considered for randomization either prior to delivery or in the first 7 hours after delivery, to accommodate the need for the first dose of study medication or placebo 8 hours after surgery. Only patients who agree to inclusion after informed consent will be randomized per protocol.

ELIGIBILITY:
Inclusion Criteria:

* Women >18 and <50 years
* BMI >30kg/m2
* Decision by clinical team to perform Cesarean section
* Rupture of membranes (ROM) < 24 hours after onset of labor or during the course of labor (ROM defined by spontaneous or artificial rupture of the amniotic sac)

Exclusion Criteria:

* Subject unwilling or unable to provide consent
* No prenatal care or a non-UTMB subject who is unlikely to be followed up after delivery
* Fetal demise or major congenital anomaly
* Immunosuppressed subjects: i.e., taking systemic immunosuppressants or steroids (e.g. transplant subjects; not including steroids for lung maturity), HIV with CD4<200, or other
* Diagnosis or suspicion of chorioamnionitis prior to randomization
* Other planned post-operative antibiotic administration
* High likelihood of additional surgical procedure beyond cesarean (e.g. scheduled hysterectomy, bowel or adnexal surgery)
* Known allergy or contraindication to cephalosporins or metronidazole
* Incarcerated individuals

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 321 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2023-07-21 (Actual); Study Completion 2023-07-21 (Actual)

PRIMARY OUTCOMES:
Surgical site infection | 6 weeks postpartum
  Including superficial or deep incisional surgical site infection, endometritis, and other related infections, such as septic pelvic thrombophlebitis and abdominal or pelvic abscess

SECONDARY OUTCOMES:
Maternal mortality | 6 weeks (42 days) postpartum
  Maternal death
Febrile morbidity | 6 weeks (42 days) postpartum
  If the patient develops a measured temperate greater than or equal to 100.4 degrees Fahrenheit (or 38.0 degrees Celsius), she will have a postpartum fever.
Postpartum antibiotic use | 6 weeks (42 days) postpartum
  We will assess via chart review and direct patient inquiry whether or not antibiotics were taken by the patient for any purpose during the six weeks (42 days) immediately following delivery.
Wound hematoma or seroma | 6 weeks (42 days) postpartum
  Wound hematoma or seroma, as diagnosed by a medical provider, according to CDC guidelines for diagnosis of wound hematoma or seroma
Use of resources | 6 weeks (42 days) postpartum
  We will note whether the patient required hospital re-admission, emergency department visits, or need for imaging or other invasive procedures
Other adverse events | 6 weeks postpartum
  Such as allergic reaction to study medications

CONTACTS AND LOCATIONS:
Overall Officials: Antonio F Saad, MD, Principal Investigator — University of Texas
Locations (2):
- United States (2):
  - St. David's North Austin Medical Center, Austin, Texas
  - University of Texas Medical Branch John Sealy Hospital, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Saad AF, Goldman B, Spencer N, Kuhlmann M, McDonnold M, Saade GR. Prophylactic Oral Cephalexin and Metronidazole Compared With Placebo After Cesarean Delivery to Reduce Infection Complications in Women With Obesity: A Randomized Controlled Trial. Obstet Gynecol. 2025 May 22;146(1):113-120. doi: 10.1097/AOG.0000000000005936. PMID 40403315